CLINICAL TRIAL: NCT02869971
Title: Prostatic Artery Embolization Versus Medical Treatment in Symptomatic Benign Prostatic Hyperplasia
Acronym: PARTEM
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Ministry of Health, France (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P150917; PHRC-15-521 (Other Grant/Funding Number: French ministry of Health); 2016-A00247-44 (Other: France: ANSM)
Record Dates: First submitted 2016-07-19; First posted 2016-08-17 (Estimated); Last update posted 2022-05-03 (Actual); Status verified 2022-04

CONDITIONS: Benign Prostatic Hyperplasia
Keywords: Prostatic artery embolization; Combined Therapy; IPSS
MeSH Terms: conditions — Prostatic Hyperplasia | interventions — Drug Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Embolization (Experimental): Prostatic Arteries Embolization
  Interventions: Device: Embosphere® (Prostatic Arteries Embolization)
- Combined Therapy (Active Comparator): Combodart® : dutasteride 0.5 mg/tamsulosin 0.4 mg per day
  Interventions: Drug: Drug therapy

INTERVENTIONS:
Device: Embosphere® (Prostatic Arteries Embolization) — Prostatic Arteries Embolization with 300-500 µm trisacryl microspheres
  Arms: Embolization
Drug: Drug therapy — Combodart (dutasteride 0.5 mg/tamsulosin 0.4 mg)
  Arms: Combined Therapy

SUMMARY:
The primary objective of this trial is to compare the 9-month effect on lower urinary tract symptoms (LUTS) of Prostatic Artery Embolization (PAE) using Embosphere® versus Standard Combined Therapy (alpha-blockers plus 5 alpha-reductase inhibitors) in patients with symptomatic BPH who failed after a first line medical treatment with alpha-blockers.

The secondary objectives of this study are to:

* Estimate the impact of the 2 strategies on benign prostatic hyperplasia specific Health Status (i.e. urinary and sexual signs and symptoms) at 3, 9, 18, and 24 months, as well as the side effects of the 2 strategies;
* Report the safety of PAE;
* Evaluate patient's adherence to medical treatment;
* Analyse the costs of each strategy and report the incremental efficiency (incremental cost utility ratio) of prostatic artery embolization compared to medical treatment.

DETAILED DESCRIPTION:
Benign Prostatic Hyperplasia (BPH) is the primary cause of lower urinary tract symptoms (LUTS) and affects > 50% of men >60 years. Moderate to severe symptoms prevalence is around 14% in France, and the proportion of men with moderate to severe symptoms doubles with each decade of age. The first-line treatment of bothersome BPH-related LUTS is medical therapy as recommended by French and European guidelines. 5α reductase inhibitors (5-ARI) can be combined with alpha-blockers and allow reduction of the size of the prostate and LUTS improvement. The severity of symptoms is usually assessed using the International prostate symptom score (IPSS) which is the standard questionnaire for the objective assessment of LUTS.

Recently, Prostatic Artery Embolization (PAE) has been proposed to treat symptomatic BPH with good safety and efficacy in single-centre studies (12-point IPSS reduction at 3 months maintained up to one year. In a randomized trial comparing PAE versus transurethral resection of prostate (TURP), Gao reported a 16-point IPSS reduction at 6 months, and an increase in the maximum urinary flow rate (Qmax) comprised between 12 ml/s and 24 ml/s at 6 months and up to 21 ml/s at 2 years. The complication rate is low (a few cases of bladder ulcer have been published) and the patient generally experiences mild post-embolization symptoms for few days.

PAE can be performed during a one-day hospitalisation and could be very attractive to patients which have insufficient benefit of medical treatment or who have side effects affecting their quality of life. The most used device for PAE is Embosphere® (Merit Medical). It bears the European CE (Conforme aux Exigences) marking for this specific indication and approximately 500 patients have been treated with it worldwide. Nonetheless, no big randomized study has proven its efficacy compared with best medical treatment. A study comparing PAE using Embosphere® and surgery (TURP) is currently enrolling patients; no patients could be included in France because men with BPH refused to be potentially assigned the surgical arm.

To properly evaluate PAE, the investigators designed the PARTEM trial, which has received the support of both the Societe Francaise de Radiologie (French society of radiology) and of the Association Francaise d'Urologie (French association of urology).

PARTEM will compare prospectively the benefit of PAE using Embosphere® to the benefit of combined medical treatment (Combodart®: Dutasteride 0.5mg Tamsulosin 0.4mg) at 9 months with an extended follow up at 24 months in order to evaluate the stability of results in both groups.

The investigators plan a multicentre, prospective, randomized, open label, parallel trial, comparing PAE to Combined Therapy (CT: alpha-blockers + 5-ARI treatment). Treatments will be allocated by minimization with a 1:1 ratio, based on study centre, IPSS score (moderate/severe) and prostate volume (< 80 g/≥80 g).

This study is designed to demonstrate the superiority of PAE to decrease LUTS compared to best medical treatment.

ELIGIBILITY:
Inclusion Criteria:

* Men aged>= 50 and <=85 years AND
* Moderate to severe LUTS defined as IPSS > 11, and QoL > 3 AND
* No improvement after an alpha blocker treatment line (Tamsulosin 0.4 mg p.d. during 1 month) AND
* Prostatic volume >=50 ml AND
* Affiliated to a French health insurance system

Exclusion Criteria:

* Severe allergy to iodine contrast agent
* Treatment with 5-ARI on the last 6 months
* Suspected prostate cancer requiring specific management
* On-going prostatitis
* On-going urinary retention
* On-going acute urinary infection
* Acontractile detrusor
* Neurogenic lower urinary tract dysfunction
* Urethral stenosis
* Bladder diverticulum
* Bladder stone with surgical indication
* Patient refusing PAE
* Creatinine clearance <40 ml/min
* Severe liver failure
* Contra-indication to alpha-blockers
* Hypersensitivity to dutasteride, other 5-alpha reductase inhibitors, tamsulosin (including case of tamsulosin induced angioedema), soya, peanut or one of the excipients
* Hypersensitivity to gelatin or collagen
* Patients ineligible for pelvic angiography
* History of orthostatic hypotension
* Patient unable or unwilling to provide written informed consent
* Patient under legal protection

Ages: 50 Years to 85 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2016-08 (Actual); Primary Completion 2020-12-03 (Actual); Study Completion 2022-03-25 (Actual)

PRIMARY OUTCOMES:
Change in IPSS score | 9 months

SECONDARY OUTCOMES:
Number of Adverse Events | 3, 9, 18, 24 months
IPSS | 3, 18, 24 months
Qmax | 3, 9, 24 months
International Index of Erectile Function (IIEF) score | 3, 9, 18, 24 months
prostate volume | 3, 9, 24 months
Prostate-Specific Antigen (PSA) level | 3, 9, 18, 24 months
Quality of life score | 3, 9, 18, 24 months
  assessed by IPSS/Quality of Life (QoL) form
Treatment units' account | 3, 9 months
  adherence to treatment
Adherence to treatment questionnaire | 3, 9 months
  adherence to treatment
number of PAE | 24 months
number of surgical treatment | 24 months
number of medication | 3, 9, 18, 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Marc Sapoval, MD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (13):
- France (13):
  - CHU de Lyon hopital Edouard Herriot, Lyon, Auvergne-Rhône-Alpes
  - CHU de Lyon centre hospitalier Lyon Sud, Pierre-Bénite, Auvergne-Rhône-Alpes
  - CHU Rennes hopital Pontchaillou, Rennes, Brittany Region
  - CHU de Bordeaux groupe hospitalier Pellegrin, Bordeaux, Nouvelle-Aquitaine
  - CHU de Limoges, Limoges, Nouvelle-Aquitaine
  - CHU Montpellier hopital Arnaud de Villeneuve, Montpellier, Occitanie
  - CHU Montpellier hopital Lapeyronie, Montpellier, Occitanie
  - AP-HM hopital la Conception, Marseille, Provence-Alpes-Côte d'Azur Region
  - AP-HM hopital de la Timone, Marseille, Provence-Alpes-Côte d'Azur Region
  - AP-HP hopital Henri-Mondor, Créteil, Île-de-France Region
  - AP-HP - Hôpital Saint-Louis, Paris, Île-de-France Region
  - AP-HP hopital Cochin, Paris, Île-de-France Region
  - AP-HP Hopital Europeen Georges Pompidou, Paris, Île-de-France Region

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Sapoval M, Thiounn N, Descazeaud A, Dean C, Ruffion A, Pagnoux G, Duarte RC, Robert G, Petitpierre F, Karsenty G, Vidal V, Murez T, Vernhet-Kovacsik H, de la Taille A, Kobeiter H, Mathieu R, Heautot JF, Droupy S, Frandon J, Barry Delongchamps N, Korb-Savoldelli V, Durand-Zaleski I, Pereira H, Chatellier G; PARTEM study group. Prostatic artery embolisation versus medical treatment in patients with benign prostatic hyperplasia (PARTEM): a randomised, multicentre, open-label, phase 3, superiority trial. Lancet Reg Health Eur. 2023 Jun 26;31:100672. doi: 10.1016/j.lanepe.2023.100672. eCollection 2023 Aug. PMID 37415648